CLINICAL TRIAL: NCT02539108
Title: Safety and Immunogenicity of the 2015-2016 Formulation of Fluzone® Quadrivalent (Influenza Vaccine) Among Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC58; U1111-1161-2526 (Other: WHO)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Fluzone® Quadrivalent Influenza Vaccine (No Preservative)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group 1 (Experimental): Participants at 6 months to < 36 months age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative
- Study Group 2 (Experimental): Participants at 3 years to < 9 years age at enrollment
  Interventions: Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative

INTERVENTIONS:
Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative — 0.25 mL, Intramuscular (Pediatric Dose, 2015 2016 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Study Group 1
Biological: Fluzone® Quadrivalent Influenza Vaccine, No Preservative — 0.5 mL, Intramuscular (2015 2016 formulation)
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Study Group 2

SUMMARY:
The study will evaluate the safety and immunogenicity of the 2015-2016 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule, in accordance with the Advisory Committee on Immunization Practices (ACIP) recommendations, in children 6 months to < 9 years of age.

Objective:

* To describe the safety of the 2015-2016 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule, in accordance with ACIP recommendations, in children 6 months to < 9 years of age.

Observational objectives:

* To describe the immunogenicity of the 2015-2016 formulation of Fluzone Quadrivalent vaccine, administered in a 1- or 2-dose schedule in accordance with ACIP recommendations, in children 6 months to < 9 years of age.
* To submit available sera from each subject to Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the FDA to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
Study participants will be assigned to the appropriate age group (6 months to < 36 months of age or 3 years to < 9 years of age) based on the subject's age at the time of enrollment. Participants aged 6 months to < 36 months will receive a 0.25 mL dose of Fluzone Quadrivalent vaccine and those aged 3 years to < 9 years will receive a 0.5 mL dose of Fluzone Quadrivalent vaccine. Participants, for whom 2 doses of influenza vaccine are recommended per ACIP guidance, will receive a second dose of Fluzone Quadrivalent vaccine during Visit 2 (28 days after Visit 1).

Solicited adverse event (AE) information will be collected for 7 days after each vaccination, unsolicited AE information will be collected from Visit 1 to Visit 2 or to Visit 3 for those subjects receiving 2 doses. Serious adverse event (SAE) information will be collected from Visit 1 to Visit 2 or Visit 3, as appropriate.

Immunogenicity will be evaluated in all subjects prior to vaccination on Day 0 (Visit 1) and at Day 28 after the final vaccination using the hemagglutination inhibition (HAI) technique. For each influenza vaccine strain, pre- and post-vaccination geometric mean titers (GMTs) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 6 months to < 9 years of age on the day of first study vaccination (study product administration)
* Subject and parent/guardian are willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study
* Assent form has been signed and dated by subjects 7 to < 9 years of age, and informed consent form has been signed and dated by parent(s) or guardian for subjects 6 months to < 9 years of age
* For subjects 6 months to < 12 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone Quadrivalent vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2 for subjects receiving 1 dose of influenza vaccine or Visit 3 for subjects receiving 2 doses of influenza vaccine
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Prior vaccination with any formulation of 2015-2016 influenza vaccine
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Identified as a natural or adopted child of the Investigator or an employee with direct involvement in the proposed study.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Bardstown, Kentucky
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 31 August 2015 to 30 November 2015 at 2 clinic centers in the United States.
Pre-assignment Details: A total of 60 participants who met all inclusion and no exclusion criteria were enrolled and vaccinated.
Groups:
- 6 to <36 Months of Age: Children 6 to <36 months of age received 1 intramuscular dose of Fluzone Quadrivalent Vaccine. A second dose was administered 28 days after the first vaccination in participants for whom a second dose was recommended according to Advisory Committee on Immunization Practices guidelines.
- 3 to <9 Years of Age: Children 3 to <9 years of age received 1 intramuscular dose of Fluzone Quadrivalent Vaccine. A second dose was administered 28 days after the first vaccination in participants for whom a second dose was recommended according to Advisory Committee on Immunization Practices guidelines.
Period: Overall Study
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.9 (8.59) | 72.0 (22.9) | 46.9 (30.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 10 | 16 | 26
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection-Site and Solicited Systemic Reactions Following Vaccination With the 2015-2016 Formulation of Fluzone® Quadrivalent Influenza Vaccine.
Description: Solicited injection-site reactions for 6 to < 36 months: Tenderness, Erythema, and Swelling. For 3 to < 9 years: Pain, Erythema, and Swelling. Solicited systemic reactions for 6 to < 36 months: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. For 3 to < 9 years: Fever (Temperature), Headache, Malaise, and Myalgia.
  Grade 3 for 6 to < 36 months: Tenderness, Cries when injected limb is moved; Erythema and Swelling, ≥ 50 mm; Vomiting, 6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal, > 3 hours; Drowsiness, sleeping most of the time or difficult to wake up; Appetite lost, Refuses ≥ 3 feeds/meals or refuses most feeds/meals; and Irritability, Inconsolable.
  Grade 3 for 3 to < 9 years: Pain, Incapacitating; Erythema and Swelling, ≥ 50 mm; Fever, ≥ 39.0°C; Headache, Malaise, and Myalgia, prevents daily activity.
Time Frame: Day 0 up to Day 7 post any vaccination
Population: Solicited injection-site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Number analyzed (Participants) | 30 | 30
Participants
  Injection-Site Tenderness (N=30, 0) | 21 | NA — Event was not assessed in this group
  Grade 3 Injection-Site Tenderness | 0 | NA — Event was not assessed in this group
  Injection-Site Pain (N=0, 30) | NA — Event was not assessed in this group | 16
  Grade 3 Injection-site Pain | NA — Event was not assessed in this group | 0
  Injection-Site Erythema | 11 | 11
  Grade 3 Injection-Site Erythema | 0 | 0
  Injection-Site Swelling | 3 | 8
  Grade 3 Injection-Site Swelling | 0 | 0
  Fever | 4 | 2
  Grade 3 Fever | 0 | 2
  Vomiting (N=30, 0) | 1 | NA — Event was not assessed in this group
  Grade 3 Vomiting | 0 | NA — Event was not assessed in this group
  Crying abnormal (N=30, 0) | 9 | NA — Event was not assessed in this group
  Grade 3 Crying abnormal | 0 | NA — Event was not assessed in this group
  Drowsiness (N=30, 0) | 8 | NA — Event was not assessed in this group
  Grade 3 Drowsiness | 0 | NA — Event was not assessed in this group
  Appetite lost (N=30, 0) | 9 | NA — Event was not assessed in this group
  Grade 3 Appetite lost | 0 | NA — Event was not assessed in this group
  Irritability (N=30, 0) | 15 | NA — Event was not assessed in this group
  Grade 3 Irritability | 0 | NA — Event was not assessed in this group
  Headache (N=0, 30) | NA — Event was not assessed in this group | 2
  Grade 3 Headache | NA — Event was not assessed in this group | 0
  Malaise(N=0, 30) | NA — Event was not assessed in this group | 6
  Grade 3 Malaise | NA — Event was not assessed in this group | 0
  Myalgia (N=0, 30) | NA — Event was not assessed in this group | 10
  Grade 3 Myalgia | NA — Event was not assessed in this group | 0

2. Secondary Outcome: Geometric Mean Titers of Influenza Virus Antibodies Following Vaccination With the 2015-2016 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay.
Time Frame: Day 0 (pre-vaccination) and 28 days post-last vaccination
Population: Anti-influenza antibody titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Number analyzed (Participants) | 30 | 30
Titers (1/dilutions)
  A/H1N1; Pre-vaccination | 14.8 [8.60 to 25.5] | 184 [85.3 to 396]
  A/H1N1; Post-vaccination | 288 [167 to 498] | 937 [625 to 1406]
  A/H3N2; Pre-vaccination | 28.9 [13.5 to 62.0] | 139 [79.8 to 243]
  A/H3N2; Post-vaccination | 1140 [576 to 2259] | 3263 [2255 to 4721]
  B Yamagata; Pre-vaccination | 16.2 [10.7 to 24.7] | 113 [64.3 to 199]
  B Yamagata; Post-vaccination | 408 [257 to 646] | 1028 [659 to 1604]
  B Victoria; Pre-vaccination | 14.0 [8.35 to 23.4] | 108 [54.1 to 216]
  B Victoria; Post-vaccination | 339 [207 to 555] | 718 [462 to 1118]

3. Secondary Outcome: Number of Participants Who Achieved Seroprotection to Influenza Virus Antigens Pre- and Post-Vaccination With the 2015-2016 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay. Seroprotection was defined as a pre-vaccination or post-vaccination influenza antibody titer of ≥ 1:40 (1/dilutions).
Time Frame: Day 0 (pre-vaccination) and 28 days post-last vaccination
Population: Anti-influenza antibody titers were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Number analyzed (Participants) | 30 | 30
Participants
  A/H1N1; Pre-vaccination | 10 | 22
  A/H1N1; Post-vaccination | 28 | 30
  A/H3N2; Pre-vaccination | 14 | 26
  A/H3N2; Post-vaccination | 29 | 30
  B Yamagata; Pre-vaccination | 8 | 23
  B Yamagata; Post-vaccination | 29 | 30
  B Victoria; Pre-vaccination | 7 | 20
  B Victoria; Post-vaccination | 28 | 30

4. Secondary Outcome: Number of Participants Who Achieved Seroconversion Following Vaccination With the 2015-2016 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition (HAI) assay. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-final vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-final vaccination titer.
Time Frame: 28 days post-last vaccination
Population: Anti-influenza antibody titers were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Number analyzed (Participants) | 30 | 30
Participants
  A/H1N1 | 24 | 15
  A/H3N2 | 28 | 28
  B Yamagata | 28 | 24
  B Victoria | 27 | 21

5. Secondary Outcome: Geometric Mean Titer Ratios of Influenza Virus Antibodies Following Vaccination With the 2015-2016 Formulation of Fluzone® Quadrivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using an hemagglutination inhibition assay. Geometric mean of titer ratio is the geometric mean of the individual post-vaccination/pre-vaccination titer ratios
Time Frame: Day 0 (pre-vaccination) and 28 days post-last vaccination
Population: Anti-influenza antibody titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Number analyzed (Participants) | 30 | 30
Titer ratio
  A/H1N1 | 13.0 [7.63 to 22.1] | 4.59 [2.93 to 7.21]
  A/H3N2 | 28.2 [17.0 to 46.8] | 22.9 [15.0 to 34.9]
  B Yamagata | 21.1 [13.5 to 32.9] | 8.67 [5.76 to 13.1]
  B Victoria | 17.3 [10.8 to 28.0] | 6.35 [4.17 to 9.66]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to 28 days following the last vaccination.
Groups:
- 6 to <36 Months of Age: Children 6 to < 36 months of age received 1 intramuscular dose of Fluzone Quadrivalent Vaccine. A second dose was administered 28 days after the first vaccination in participants for whom a second dose was recommended according to Advisory Committee on Immunization Practices guidelines.
- 3 to <9 Years of Age: Children 3 to < 9 years of age received 1 intramuscular dose of Fluzone Quadrivalent Vaccine. A second dose was administered 28 days after the first vaccination in participants for whom a second dose was recommended according to Advisory Committee on Immunization Practices guidelines.
Arm/Group | 6 to <36 Months of Age | 3 to <9 Years of Age
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 21/30 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 to <36 Months of Age (N=30) | 3 to <9 Years of Age (N=30)
Linear IgA disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 to <36 Months of Age (N=30) | 3 to <9 Years of Age (N=30)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Teething (Gastrointestinal disorders) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Injection site Tenderness / Pain (General disorders) | 21 (21) | 16 (16)
Injection site Erythema (General disorders) | 11 (11) | 11 (11)
Injection site Swelling (General disorders) | 3 (3) | 8 (8)
Fever (General disorders) | 4 (4) | 2 (2)
Crying abnormal (Psychiatric disorders) | 9 (9) | 0 (0)
Drowsiness (Nervous system disorders) | 8 (8) | 0 (0)
Appetite lost (Metabolism and nutrition disorders) | 9 (9) | 0 (0)
Irritability (Psychiatric disorders) | 15 (15) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications